CLINICAL TRIAL: NCT04221841
Title: University of Bojnord
Brief Title: Executive Functions and Reinforcement Sensitivity in Women With Obsessive Compulsive Symptoms
Status: Completed | Type: Observational
Sponsor: Malahat Amani (Other)
Responsible Party: Sponsor-Investigator, Malahat Amani, assistant professor, University of Bojnord
Organization: University of Bojnord (Other)
Other Study IDs: 131820
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Obsessive-Compulsive Symptom; Executive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: descriptive — correlation

SUMMARY:
Methods: The study population consisted of all adult women living in Sabzevar city (Iran). Using cluster sampling, 365 women were selected as the study sample. Participants completed Obsessive-Compulsive Inventory, Sensitivity to Punishment and Sensitivity to Reward Questionnaire - Revised and Clarified (SPSRQ-RC) as well as Behavior Rating Inventory of Executive Function (BRIEF). Data analysis was conducted using correlation and regression tests.

ELIGIBILITY:
Inclusion Criteria:

having age between 18 to 54, be female, be literacy,

Exclusion Criteria:

be male, be illiteracy, having psychotic disorders

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The statistical population consisted of all adult women living in Sabzevar city in 2019. The sampling was conducted using cluster sampling method. In randomly selected areas, participants were selected from among local women
Sampling Method: Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
executive functions | 1 month
  It was measured by behavior rating inventory of executive function. it consists of 75 items that are measured on a 5-point Likert scale. subscales include inhibition, shift, emotional control, self-monitoring, initiation, working memory, planning/organization, task monitoring and organization of materials. min and max scores are 0 and 150. respectively. the higher scores indicate problems in executive functions.
obsessive-compulsive symptom | 1 month
  it was measured by the Obsessive-Compulsive Inventory. This inventory contains 42 items that are measured on a 5-point Likert scale. It consists of the sub-scales of washing, controlling, doubting, ordering, obsession, hoarding, and neutralizing. the higher scores are probably an indicator of obsessive-compulsive disorder.
reinforcement sensitivity | 1 month
  it was measured by Sensitivity to Punishment and Sensitivity to Reward Questionnaire: This 20-item scale measures sensitivity to reward and sensitivity to punishment, which is scored on a 5-point Likert scale (from "totally correct" to "totally incorrect"). the higher scores in subscales of sensitivity to punishment and Sensitivity to Reward indicate high activity in punishment and reward systems.

CONTACTS AND LOCATIONS:
Locations (1):
- Malahat Amani, Bojnourd, North Khorasan, Iran